CLINICAL TRIAL: NCT02109679
Title: Relative Bioavailability of Multiple Oral Doses of BI 187004 and Metformin After Co-administration Compared to Multiple Oral Doses of BI 187004 Alone and Metformin Alone in Healthy Male Subjects (an Open-label, Randomised, Two-sequence Crossover Study)
Brief Title: Relative Bioavailability of Multiple Oral Doses of BI 187004 and Metformin After Co-administration Compared to Multiple Oral Doses of BI 187004 Alone and Metformin Alone in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1307.7; 2013-004628-13 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin

ARMS (3):
- Treatment A (Experimental): multiple doses BI 187004
  Interventions: Drug: BI 187004
- Treatment B (Experimental): multiple doses BI 187004 + multiple doses metformin
  Interventions: Drug: BI 187004; Drug: metformin
- Treatment C (Experimental): multiple doses metformin
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: metformin — multiple doses metformin given as tablet
  Arms: Treatment C
Drug: BI 187004 — multiple doses BI 187004 given as tablets
  Arms: Treatment A
Drug: BI 187004 — multiple doses BI 187004 given as tablets
  Arms: Treatment B
Drug: metformin — multiple doses metformin given as tablet
  Arms: Treatment B

SUMMARY:
To investigate bioavailability of BI 187004 and of metformin after concomitant multiple oral administration of 240 mg BI 187004 q.d. and 1000 mg metformin b.i.d. in comparison to BI 187004 and metformin given alone.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects
2. Subjects must be able to understand and comply with study requirements
3. Age of 18 to 50 years
4. Body mass index (BMI) of 18.5 to 29.9 kg/m2

Exclusion criteria:

1. Any finding in the medical examination (including BP, pulse rate (PR) or ECG) is deviating from normal and judged as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg or diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease judged as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication (except appendectomy and simple hernia repair)
7. Diseases of the central nervous system (such as epilepsy), other neurological disorders or psychiatric disorders

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
AUCt,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval t) for BI 187004 | up to 24 hours postdose
AUCt,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval t) for metformin | up to 12 hours postdose
Cmax,ss (Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval t) for BI 187004 | up to 24 hours postdose
Cmax,ss (Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval t) for metformin | up to 12 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1307.7.1 Boehringer Ingelheim Investigational Site, Biberach, Germany